CLINICAL TRIAL: NCT06848010
Title: TRacheal Cuff PRessure Evaluation Study
Acronym: TRAC-PRES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Giacomo Grasselli, Prof, Policlinico Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TRAC-PRES
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pneumonia, Ventilator-Associated; Mechanical Ventilation
Keywords: pressure cuff control; mechanical ventilation
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automated endotracheal cuff controller (Experimental): The endotracheal tube cuff pressure will be continuously controlled by the Trachflush system, at pre-specifed pressure level of 25 cmH20.
  Interventions: Device: Automated endotracheal cuff controller
- Control group (analogic manometer) (No Intervention): The endotracheal cuff will be inflated at 25 cmH20 manually by an analogic manometer. Every 8 hours analogic manometry will be performed to assess cuff pressure.

INTERVENTIONS:
Device: Automated endotracheal cuff controller — The automated endotracheal tube cuff pressure controller will continously assess and maintain the endotracheal tube cuff pressure at pre-specifed pressure level of 25 cmH20.
  Arms: Automated endotracheal cuff controller

SUMMARY:
Randomized clinical trial in mechanically ventilate critically ill patients. The study will evaluated the efficacy of a continous endotracheal tube (ETT) cuff pressure controller (TRACH FLUSH group) compared to manual monitoring and inflation (STANDARD group).

Patients intubated, from at least 24 hours and with a predicted duration of invasive mechanical ventilation longer than 72 hours, will be randomized to the use of TRACH FLUSH versus nurse operated analogic cuff pressure controller q8.

Hypotesis of the study is the superiority of the continuous cuff pressure controller in maintaining cuff pressure within the target value, thus decreasing the incidence of microaspiration events.

Aim of the study are 1) to compare the incidence of cuff pressure value detection outside the target range between the TRACH FLUSH and the STANDARD group, and 2) to compare the incidence of sputum samples positive for (amylase and/or pepsin), a surrogate for tracheal micro-aspiration event.

DETAILED DESCRIPTION:
Endotracheal intubation is an effective method of providing rapid and safe airway patency and respiratory support in the intensive care unit (ICU). Endotracheal intubation effectively isolates the trachea by inflating the endotracheal tube (ETT) cuff just below the vocal cords: this ensures airway patency and positive pressure ventilation. The pressure of the endotracheal tube cuff (Pcuff) should be between 20-30 cmH2O to ensure airway isolation. The literature reports that overinflation of the endotracheal cuff (>30 cmH2O) causes hoarseness, sore throat, inadequate swallowing of secretions, tracheal stenosis, tracheal wall damage, and ischemia due to decreased mucosal capillary blood flow: these changes can occur even if a high Pcuff is maintained for a short period of time. In contrast, inadequate inflation (less than 20 cmH2O) results in ventilation-associated pneumonia (VAP) due to ineffective ventilation and microaspiration of gastric and/or oropharyngeal secretions into the lungs. Risk factors for microaspiration include patient-related factors, factors related to endotracheal tube type, performance of invasive procedures such as enteral nutrition through a nasogastric or orogastric tube, and mechanical ventilation. Patient-related factors include supine position, sedation, coma, tracheal diameter, and viscosity of secretions, while among those related to tube type we find impossible vocal cord closure, longitudinal folds of low-pressure and high-volume polyvinyl chloride (PVC) tracheal tubes. The American Association of Critical-Care Nurses (AACN) states that in order to achieve adequate pressure and prevent mucosal damage, the amount of pressure and volume of air needed, the size, shape of the tube, mode of mechanical ventilation, and the patient's blood pressure must be taken into account.

The methods found in ICUs to control Pcuff and keep it within safe ranges are about a dozen and range from manual external palpation of the inflation balloon, to assessment of inspiratory/expiratory volume loss to continuous monitoring with appropriate instrumentation.

Despite the known Pcuff-related complications of ETT, there is a paucity of national or international guidelines on the optimal pressure value, frequency of pressure measurement, and measurement methods: however, some studies performed show that the use of an automated device that continuously monitors Pcuff significantly decreases gastric microaspirations.

ELIGIBILITY:
Inclusion Criteria:

* Required invasive mechanical ventilation expected to last for more than 24h
* Signed informed consent

Exclusion Criteria:

* Intubated from more than 6 hours at the time of screening
* Pregnancy
* Previous surgery involving the airways

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cuff Pressure | From enrollment to either the 5th day of invasive mechanical ventilation, or discontinuation of invasive mechanical ventilation
  Incidence of measurements with a endotracheal cuff pressure outside the prespecified target value: 25 cmH2O

SECONDARY OUTCOMES:
Microaspiration | From enrollment to either the 5th day of invasive mechanical ventilation, or discontinuation of invasive mechanical ventilation
  Incidence of detection of detectable levels of Pepsin A and Amylase in the tracheal secretions samples. Daily sampling of tracheal secretions will be performed at 8:00AM.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Zanella, MD, Study Chair — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data regarding characteristics of patients enrolled, treatment performed and outcome will be available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the completion of patients enrollement and once study data have been verified by investigators. Data will be available for undefinite time.
Access Criteria: Researchers interested in the topic, previous authorization of the principal investigator

REFERENCES:
- [Background] Kumar CM, Seet E, Van Zundert TCRV. Measuring endotracheal tube intracuff pressure: no room for complacency. J Clin Monit Comput. 2021 Feb;35(1):3-10. doi: 10.1007/s10877-020-00501-2. Epub 2020 Mar 20. PMID 32198671
- [Background] Hamilton VA, Grap MJ. The role of the endotracheal tube cuff in microaspiration. Heart Lung. 2012 Mar-Apr;41(2):167-72. doi: 10.1016/j.hrtlng.2011.09.001. Epub 2011 Dec 30. PMID 22209048
- [Background] Blot SI, Poelaert J, Kollef M. How to avoid microaspiration? A key element for the prevention of ventilator-associated pneumonia in intubated ICU patients. BMC Infect Dis. 2014 Nov 28;14:119. doi: 10.1186/1471-2334-14-119. PMID 25430629